CLINICAL TRIAL: NCT01986920
Title: A Randomized, Double-Blind, Vehicle-Controlled, Within-Subject, Comparison Study of the Safety, Tolerability, And Effectiveness of A-101 Topical Solution in Subjects With Seborrheic Keratosis
Brief Title: Study of Safety, Tolerability and Effectiveness of A-101 in Subjects With Seborrheic Keratosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-101-SEBK-201
Record Dates: First submitted 2013-11-06; First posted 2013-11-19 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Seborrheic Keratosis (SK)
Keywords: SK; Seborrheic Keratosis
MeSH Terms: conditions — Keratosis, Seborrheic | interventions — N-phenylacetoaminomethylene-DL-p-nitrophenylalanine

STUDY DESIGN:
Intervention Model Description: The three tests solutions and the placebo solution are each applied topically to 1 of 4 target lesions on the backs of each subject (determined by the randomization schedule). If needed a second treatment may be applied at Visit 5.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A-101 25% (Active Comparator): Low dose group
  Interventions: Drug: A-101 25%
- A-101 32.5% (Active Comparator): Mid Dose Group
  Interventions: Drug: A-101 32.5%
- A-101 40% (Active Comparator): High Dose Group
  Interventions: Drug: A-101 40%
- A-101 Vehicle (Placebo Comparator): Placebo group
  Interventions: Drug: A-101 Vehicle

INTERVENTIONS:
Drug: A-101 25% — Low Dose Concentration of A-101 applied to one of 4 Target Lesions
  Arms: A-101 25%
Drug: A-101 32.5% — Mid Dose Concentration of A-101 applied to one of 4 Target Lesions
  Arms: A-101 32.5%
Drug: A-101 40% — High Dose Concentration A-101 applied to one of 4 Target Lesions
  Arms: A-101 40%
Drug: A-101 Vehicle — Placebo applied to one of 4 Target Lesions
  Arms: A-101 Vehicle

SUMMARY:
Evaluate the safety, tolerability of A-101 when applied to seborrheic keratosis lesions on the back of subjects.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the safety, effectiveness and tolerability of three concentrations of A-101 25%, 32.5%, and 40%, when applied to individual seborrheic keratosis target lesions on the back compared with a matching A-101 vehicle.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age
2. Has a clinical diagnosis of stable clinically typical seborrheic keratosis
3. Has at least 4 appropriate seborrheic keratosis target lesions on the back
4. If subject is a women of childbearing potential, she must have a negative urine pregnancy test and must agree to use an active form of birth control for the duration of the study
5. Is non-pregnant and non-lactating
6. Is in good general health and free of any disease state or physical condition which, in the investigator's opinion, might impair evaluation of any target lesion or which exposes the subject to an unacceptable risk by study participation
7. Is willing and able to follow all study instructions and to attend all study visits
8. Is able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. Has clinically atypical and/or rapidly growing seborrheic keratosis lesions
2. Has presence of multiple eruptive seborrheic keratosis lesions (Sign of Leser-Trelat)
3. Has used any of the following systemic therapies within the specified period prior to Visit 1:

   * Retinoids; 180 days
   * Glucocorticosteroids; 28 days
   * Anti-metabolites (e.g., methotrexate); 28 days
4. Has used any of the following topical therapies on the treatment area within the specified period prior to Visit 1:

   * Retinoids; 90 days
   * Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-fluorouracil, or ingenol mebutate; 60 days
   * Glucocorticosteroids or antibiotics; 14 days
   * Moisturizers/emollients, sunscreens; 12 hours
5. Has had any LASER, light (e.g., intense pulsed light (IPL), photo-dynamic therapy (PDT)) or other energy based therapy on the treatment area within 180 days prior to Visit 1
6. Has a history of keloid formation or hypertrophic scarring
7. Has a current systemic malignancy
8. Has a history of, within the 180 days prior to Visit 1, or has a current cutaneous malignancy on the treatment area
9. Has a current pre-malignancy (e.g., actinic keratosis) on the treatment area
10. Has had body art (e.g., tattoos, piercing, sculpting, etc.) or any other invasive, non-therapeutic procedure performed on the treatment area that, in the opinion of the investigator, might put the subject at undue risk or interfere with the study conduct or evaluations
11. Has excessive tan on the treatment area that, in the opinion of the investigator, might put the subject at undue risk or interfere with the study conduct or evaluations
12. Has experienced a sunburn on the treatment area within the previous 4 weeks
13. Has a history of sensitivity to any of the ingredients in the study medications
14. Has any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or condition (e.g., sunburn, tattoos, excessive hair, open wounds on the back) that, in the opinion of the investigator, might put the subject at undue risk or interfere with the study conduct or evaluations
15. Has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-10-22; Primary Completion 2014-02-25 (Actual); Study Completion 2014-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Dubois, MD, Principal Investigator — Derm Research, PLLC
Locations (1):
- DermResearch, Inc., Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Sponsor Website — http://www.aclaristx.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study each patient is treated with all 4 treatments on 4 different lesions on their back. Therefore, each patient participates in each group so the total enrollment matches the number of lesions treated but not the total participants.
Units Other Than Participants: lesions
Period: A- 101 25%
Arm/Group | A-101 25% | A-101 32.5% | A-101 40% | A-101 Vehicle
Started (It is the same 35 participants in each treatment so total participants is 35.) | 35; 35 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Completed (Participants receives all treatments, one treatment/lesion simultaneously. 1 Participant=4 lesion) | 34; 34 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Not Completed | 1; 1 lesions | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: A-101 32.5%
Arm/Group | A-101 25% | A-101 32.5% | A-101 40% | A-101 Vehicle
Started | 0; 0 lesions | 35; 35 lesions | 0; 0 lesions | 0; 0 lesions
Completed | 0; 0 lesions | 34; 34 lesions | 0; 0 lesions | 0; 0 lesions
Not Completed | 0; 0 lesions | 1; 1 lesions | 0; 0 lesions | 0; 0 lesions
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: A-101 40%
Arm/Group | A-101 25% | A-101 32.5% | A-101 40% | A-101 Vehicle
Started | 0; 0 lesions | 0; 0 lesions | 35; 35 lesions | 0; 0 lesions
Completed | 0; 0 lesions | 0; 0 lesions | 34; 34 lesions | 0; 0 lesions
Not Completed | 0; 0 lesions | 0; 0 lesions | 1; 1 lesions | 0; 0 lesions
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Placebo
Arm/Group | A-101 25% | A-101 32.5% | A-101 40% | A-101 Vehicle
Started | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 35; 35 lesions
Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 34; 34 lesions
Not Completed | 0; 0 lesions | 0; 0 lesions | 0; 0 lesions | 1; 1 lesions
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Subjects were required to have 4 Target Seborrheic Keratosis Lesions their back. Each lesion was treated with one of the four treatment interventions (A-101 Solution 25%, A-101, Solution 32.5%, A-101 Solution 40% and the A-101 Solution Vehicle) in a randomized fashion.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.43 (6.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Physician Lesion Assessment Scale
Description: Mean Change in Score on the Physician Lesion Assessment Scale (PLA) of each Target Lesion. The PLAS is a four point scale from 0-3 with 0 being clear and 3 being the worst lesion.
  The primary effectiveness will consist of the mean change from Visit 2 to Visit 9 in PLA performed using Analysis of Covariance (ANCOVA) with Visit 2 PLAS as the covariate. Comparisons between vehicle and each active treatment group will be performed within the model using least-squares means and the common error term.
Time Frame: Visit 2 to visit 9 (78 days)
Population: A total of 35 subjects were enrolled with 34 subjects in the analysis population. Each target lesion on a subject was treated with one of the 4 study medications in a random fashion.
Measure: Mean (Standard Deviation); unit: Change in Score on a scale
Arm/Group | A-101 25% | A-101 32.5% | A-101 40% | A-101 Vehicle
Number analyzed (Participants) | 34 | 34 | 34 | 34
Change in Score on a scale | -0.47 (0.66) | -0.88 (0.73) | -1.12 (0.81) | -0.15 (0.36)

2. Secondary Outcome: Subject's Self Assessment Scale
Description: Subjects self assessment of the condition of their lesions based on a scale of Clear (Grade 0), Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3).
Time Frame: Visit 9 (Day 78)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A-101 25% | A-101 32.5% | A-101 40% | A-101 Vehicle
Number analyzed (Participants) | 34 | 34 | 34 | 34
Participants
  Clear | 7 | 09 | 08 | 01
  Mild | 12 | 09 | 13 | 13
  Moderate | 13 | 12 | 11 | 18
  Severe | 02 | 04 | 02 | 02

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time the subject signed the informed consent until the subject's last visit. Adverse events were collected from the time immediately after the first application of the study medication until the subject's last visit.
Arm/Group | A-101 25% | A-101 32.5% | A-101 40% | A-101 Vehicle
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/35 | 1/35 | 1/35
Other Adverse Events (participants affected / at risk) | 21/35 | 21/35 | 25/35 | 25/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 25% (N=35) | A-101 32.5% (N=35) | A-101 40% (N=35) | A-101 Vehicle (N=35)
Acute Pyelonephritis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A-101 25% (N=35) | A-101 32.5% (N=35) | A-101 40% (N=35) | A-101 Vehicle (N=35)
Crusting (Skin and subcutaneous tissue disorders) | 6 | 12 | 15 | 0
Erythema (Skin and subcutaneous tissue disorders) | 8 | 17 | 19 | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Hypopigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Induration (Skin and subcutaneous tissue disorders) | 3 | 4 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Scaling (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 0
Stinging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Seasonal allergy (Immune system disorders) | 10 | 10 | 10 | 10
Wound (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 4 | 4
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 1 | 1 | 1
Insomnia (Nervous system disorders) | 1 | 1 | 1 | 1
Depression (Psychiatric disorders) | 1 | 1 | 1 | 1
Cystitis (Renal and urinary disorders) | 1 | 1 | 1 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1

LIMITATIONS AND CAVEATS:
Since each patient simultaneously participates in all four treatment groups only skin site related adverse events are reported by treatment group. Systemic adverse events are reported in all treatment groups the same.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and the investigator agree not to publish the results of this study without the written approval of the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT01986920/Prot_SAP_000.pdf